CLINICAL TRIAL: NCT01240161
Title: Personalized Translational Platform for Biomarker Discovery in Brain Tumors
Status: Completed | Type: Observational
Sponsor: Marcelo F. Di Carli, MD, FACC (Other)
Collaborators: Society of Nuclear Medicine and Molecular Imaging (Unknown); General Electric (Industry)
Responsible Party: Sponsor-Investigator, Marcelo F. Di Carli, MD, FACC, Chief of Nuclear Medicine/PET, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Other Study IDs: 2008P000554
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: High Grade Glioma
Keywords: Glioblastoma multiforme; FLT; PET
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with high grade gliomas: All subjects will have radiographically suspected or surgically proven de novo high grade gliomas. There are no control patients.
  Interventions: Drug: FLT-PET/CT: (3'deoxy-3'-[(18)F] fluorothymidine) PET/CT

INTERVENTIONS:
Drug: FLT-PET/CT: (3'deoxy-3'-[(18)F] fluorothymidine) PET/CT — Each patient will have 0-3 or more FLT-PET brain scans.

SUMMARY:
The central hypothesis for this proposal is that multimodal (clinical, imaging, tissue) biomarkers will better predict early brain tumor response to treatments and will be more reliable prognostic markers in patients with malignant brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or suspected high grade glioma ≥ 1cm in diameter on postoperative anatomic imaging (contrast MRI), prior to initiation of chemoXRT
* Anticipated survival ≥6 months
* Able to give informed consent
* Capable of undergoing MRI and PET scans without the need for sedation or general anesthesia
* Male or Female

Exclusion Criteria:

* Prior radiation therapy and chemotherapy to the brain
* Active intracranial infection or nonglial brain mass.
* Recent large intracranial hemorrhage (<1 month)
* Expected survival <6 months
* Pregnant or nursing
* Renal failure
* Lives far from BWH and/or is unwilling/ unable to return for scheduled imaging visits.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to BWH/DFCI emergency department (ED), inpatient, or neurology/ neurosurgery/ radiation oncology clinics with newly diagnosed brain masses (suspected high grade gliomas) will be consented and enrolled in this study after adequate explanation of the risks and benefits of the study.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 7 months
Progression free Survival | 7 months
  MRI and clinical criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marie Kijewski, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - University of California at San Diego, San Diego, California
  - Brigham and Women's Hospital, Boston, Massachusetts